CLINICAL TRIAL: NCT02151747
Title: Pilot Study of Validation of Testing BRCA 1/2 Mutation Using Next Generation Sequencing
Brief Title: Testing BRCA 1/2 Mutation Using Next Generation Sequencing
Acronym: BRCANGS
Status: Completed | Type: Observational
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Hyung Seok Park, MD, PhD, Clinical Assistant Professor, Severance Hospital
Other Study IDs: 4-2013-0889
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Breast Neoplasms; Breast Cancer
Keywords: breast neoplasms, BRCA1, Sanger, NGS, Next generation sequencing
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sanger: BRCA 1/2 test results by Sanger sequencing
- NGS: BRCA 1/2 test results by NGS

SUMMARY:
Testing BRCA 1/2 mutation is important for patients with breast cancer, and Sanger sequencing is a standard method to identify BRCA 1/2 mutation. Next generation sequencing (NGS) is a high-throughput parallel sequencing that can provide genetic information with high accuracy. NGS is a faster and cost-effective method to detect gene mutations compared to Sanger sequencing. In this study, we evaluated the clinical role of NGS testing for BRCA 1/2 compared to Sanger sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Breast or ovarian cancer history in 2nd degree family members
* Male breast cancer
* Bilateral breast cancer
* Patient with breast cancer under 40 year of age
* Simultaneous breast and ovarian cancer
* Patients with epithelial ovarian cancer
* Breast cancer with other simultaneous extramammary malignancy

Exclusion Criteria:

-Patients who do not agree with testing BRCA 1/2 mutation

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Overall Accuracy | 1 year
  after enrollment, comparison between Sanger and NGS method will be performed.

SECONDARY OUTCOMES:
Sensitivity, Specificity | 1 year
  Sensitivity and specificity of NGS

OTHER OUTCOMES:
False negative and false positive rates | 1 year
  False negative and false positive rates of NGS

CONTACTS AND LOCATIONS:
Overall Officials: Seung IL Kim, MD, phD, Study Director — Yonsei University; JH Sohn, MD,phD, Study Director — Yonsei University; Hyung Seok Park, MD, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea